CLINICAL TRIAL: NCT04311814
Title: Valsalva Urethral Profile (VUP) : a New Measure to Assess Stress Urinary Incontinence in Women
Brief Title: The Valsalva Urethral Profile : a Measure to Assess Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poissy-Saint Germain Hospital (Other)
Responsible Party: Principal Investigator, Anne Cecile Pizzoferrato, MD, Poissy-Saint Germain Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A01411-48
Record Dates: First submitted 2020-02-21; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence; Urodynamics; Maximal urethral cloture pressure; Bladder neck mobility
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: We conducted a monocentric interventional study, carried out as part of routine care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- v-MUCP value (Other): All patients referred for urodynamics explorations will have a measure of the MUCP during a Valsalva manoeuver
  Interventions: Diagnostic Test: Maximum urethral closure pressure during Valsalva (v-MUCP)

INTERVENTIONS:
Diagnostic Test: Maximum urethral closure pressure during Valsalva (v-MUCP) — v-MUCP measurement was performed for all patients referred for urodynamic exploration of the lower urinary tract

SUMMARY:
Clinical and paraclinical appraisal of stress urinary incontinence (SUI) is mainly based on the assessment of pelvic floor muscles (PFM) contraction and urethral mobility, the measurement of the maximum urethral closure pressure (MUCP) at rest by urethral pressure profilometry (UPP) and the measurement of the Valsalva leak point pressure (VLPP).

Currently, MUCP and VLPP cannot be used for diagnosing SUI because they appear to be moderately correlated with the severity of SUI.

The lack of a specific SUI biomarker could be the explanation for the poor predictive value of urodynamics and the ongoing debate on whether urodynamic testing before surgery has benefits. Our main objective was to study the value of a new urodynamic parameter in the diagnosis of female SUI: the Valsalva urethral profile (VUP)

ELIGIBILITY:
Inclusion Criteria:

* women over the age of 18 years, referred for urodynamic exploration of the lower urinary tract, with or without lower urinary tract disorders (TUBA)
* women who gave their consent to participate in the study.

Exclusion Criteria:

* pelvic organ prolapse (POP) ≥ stage 2 according to the POP-Q classification
* history of surgery for SUI and / or POP,
* acute urinary tract infection,
* proven neurological pathology,
* urine retention,
* a history of pneumothorax
* a lability of MUCP ≥ 15 cmH2O

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Correlation between v-MUCP and diagnosis of SUI | through study completion, an average of 6 months
  Spearman correlation between the v-MCUP value and the ICIQ score. The ICIQ score (International Consultation on Incontinence Questionnaire-Urinary Incontinence) is a validated score used to quantify urinary incontinence (ranging from 0 = no incontinence to 21 = severe incontinence). v-MUCP (Valsalva Maximal Urethral Closure Pressure) is a urodynamic measure (measured in cmH2O). The Spearman correlation coefficient assesses how well the relationship between two variables can be described using a monotonic function.
Correlation between v-MUCP and MUCP | through study completion, an average of 6 months
  Spearman correlation coefficient. The Spearman correlation coefficient assesses how well the relationship between two variables can be described using a monotonic function. v-MUCP (Valsalva Maximal Urethral Closure Pressure) and MUCP Maximal Urethral Closure Pressure are two urodynamics measures (cmH2O)
Correlation between v-MUCP and VLPP | through study completion, an average of 6 months
  Spearman correlation, v-MUCP (valsalva Maximal Urethral Closure Pressure, cmH2O) and VLPP (Valsalva Leak Point Pressure, cmH2O) are urodyamic measures
Discrimination capacity of v-MUCP (valsalva Maximal Urethral Closure Pressure, cmH2O) for the diagnosis of SUI (ICIQ = 0 versus ICIQ > 0) | through study completion, an average of 6 months
  ROC curve. A Receiver Operating Characteristic (ROC) Curve is a way to compare diagnostic tests. It is a plot of the true positive rate against the false positive rate

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Dompeyre, MD, Principal Investigator — Intercommunal Hsopital center of Poissy Saint Germain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petros PE, Ulmsten UI. An integral theory and its method for the diagnosis and management of female urinary incontinence. Scand J Urol Nephrol Suppl. 1993;153:1-93. No abstract available. PMID 8108659
- [Background] DeLancey JO. Structural support of the urethra as it relates to stress urinary incontinence: the hammock hypothesis. Am J Obstet Gynecol. 1994 Jun;170(6):1713-20; discussion 1720-3. doi: 10.1016/s0002-9378(94)70346-9. PMID 8203431
- [Background] DeLancey JO, Trowbridge ER, Miller JM, Morgan DM, Guire K, Fenner DE, Weadock WJ, Ashton-Miller JA. Stress urinary incontinence: relative importance of urethral support and urethral closure pressure. J Urol. 2008 Jun;179(6):2286-90; discussion 2290. doi: 10.1016/j.juro.2008.01.098. Epub 2008 Apr 18. PMID 18423707
- [Background] Bump RC, Elser DM, Theofrastous JP, McClish DK. Valsalva leak point pressures in women with genuine stress incontinence: reproducibility, effect of catheter caliber, and correlations with other measures of urethral resistance. Continence Program for Women Research Group. Am J Obstet Gynecol. 1995 Aug;173(2):551-7. doi: 10.1016/0002-9378(95)90281-3. PMID 7645634
- [Background] McGuire EJ, Fitzpatrick CC, Wan J, Bloom D, Sanvordenker J, Ritchey M, Gormley EA. Clinical assessment of urethral sphincter function. J Urol. 1993 Nov;150(5 Pt 1):1452-4. doi: 10.1016/s0022-5347(17)35806-8. PMID 8411422
- [Background] Theofrastous JP, Bump RC, Elser DM, Wyman JF, McClish DK. Correlation of urodynamic measures of urethral resistance with clinical measures of incontinence severity in women with pure genuine stress incontinence. The Continence Program for Women Research Group. Am J Obstet Gynecol. 1995 Aug;173(2):407-12; discussion 412-4. doi: 10.1016/0002-9378(95)90260-0. PMID 7645615
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] Kirschner-Hermanns R, Anding R, Rosier P, Birder L, Andersson KE, Djurhuus JC. Fundamentals and clinical perspective of urethral sphincter instability as a contributing factor in patients with lower urinary tract dysfunction--ICI-RS 2014. Neurourol Urodyn. 2016 Feb;35(2):318-23. doi: 10.1002/nau.22815. PMID 26872575
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Messelink B, Benson T, Berghmans B, Bo K, Corcos J, Fowler C, Laycock J, Lim PH, van Lunsen R, a Nijeholt GL, Pemberton J, Wang A, Watier A, Van Kerrebroeck P. Standardization of terminology of pelvic floor muscle function and dysfunction: report from the pelvic floor clinical assessment group of the International Continence Society. Neurourol Urodyn. 2005;24(4):374-80. doi: 10.1002/nau.20144. No abstract available. PMID 15977259
- [Background] Fritel X, Fauconnier A, Bader G, Cosson M, Debodinance P, Deffieux X, Denys P, Dompeyre P, Faltin D, Fatton B, Haab F, Hermieux JF, Kerdraon J, Mares P, Mellier G, Michel-Laaengh N, Nadeau C, Robain G, de Tayrac R, Jacquetin B; French College of Gynaecologists and Obstetricians. Diagnosis and management of adult female stress urinary incontinence: guidelines for clinical practice from the French College of Gynaecologists and Obstetricians. Eur J Obstet Gynecol Reprod Biol. 2010 Jul;151(1):14-9. doi: 10.1016/j.ejogrb.2010.02.041. Epub 2010 Mar 16. PMID 20236751
- [Background] Nager CW, Schulz JA, Stanton SL, Monga A. Correlation of urethral closure pressure, leak-point pressure and incontinence severity measures. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(6):395-400. doi: 10.1007/s001920170020. PMID 11795644
- [Background] Pizzoferrato AC, Fauconnier A, Fritel X, Bader G, Dompeyre P. Urethral Closure Pressure at Stress: A Predictive Measure for the Diagnosis and Severity of Urinary Incontinence in Women. Int Neurourol J. 2017 Jun;21(2):121-127. doi: 10.5213/inj.1732686.343. Epub 2017 Jun 21. PMID 28673060
- [Background] Dietz HP, Clarke B. The urethral pressure profile and ultrasound imaging of the lower urinary tract. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(1):38-41. doi: 10.1007/s001920170092. PMID 11294530